CLINICAL TRIAL: NCT01761318
Title: Magnetic Resonance Assessment of Victoza Efficacy in the Regression of Cardiovascular Dysfunction In Type 2 Diabetes Mellitus
Brief Title: Effect of Liraglutide on Cardiovascular Endpoints in Diabetes Mellitus Type 2 Patients
Acronym: MAGNA VICTORIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, M.B. Bizino, MD, principal investigator, M.B. Bizino, MD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 379; 2012-001623-12 (EudraCT Number)
Record Dates: First submitted 2012-12-20; First posted 2013-01-04 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus Type 2; Metabolic Syndrome; Cardiovascular Disease; Diastolic Dysfunction; Fatty Liver
Keywords: Diabetes mellitus type 2; Glucagon-Like Peptide 1; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Steatosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Cardiovascular Diseases; Fatty Liver | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Active Comparator): Liraglutide: Solution for subcutaneous injection 6 mg/ml; Flexpen 3 ml.
  Dose: s.c. 0,6 mg (0,1 mL) once daily. After 1 week, the dose will be increased to 1,2 mg (0,2 mL) once daily. If tolerated, after 1 week, dose will be increased to 1.8 mg (0,3 mL) once daily. In case of a hypoglycaemic episode, the dosage of oral blood glucose lowering medicaments will be adjusted first. If hypoglycaemia persists, Liraglutide / Liraglutide placebo will be adjusted on the basis of clinical parameters.
  Duration: 26 weeks
  Interventions: Drug: Liraglutide
- Liraglutide-placebo (Placebo Comparator): Liraglutide placebo: Solution for injection; Flexpen 3 ml.
  Dosage: same as Liraglutide
  Duration: 26 weeks
  Interventions: Drug: Liraglutide - Placebo

INTERVENTIONS:
Drug: Liraglutide — Preparation and labelling of Investigational Medicinal Product:
  Liraglutide will be packed and labeled by Novo Nordisk A/S and provided in non-subject specific boxes. Labeling will be in accordance with Annex 13, local law and trial requirements. The examples of labels are not readily available, but will be supplied when received from Novo Nordisk.
  Drug accountability:
  Drug accountability will be cared for by the Department of Clinical Pharmacy of the LUMC. The trial product will be dispensed to each subject as required according to treatment group by the clinical pharmacist. No trial product will be dispensed to any person not enrolled in the trial.
  Other Names: Trade name: Victoza; EV Product Code: SUB25238; Name of the Marketing Authorisation Holder: Novo Nordisk; Marketing Authorisation number: EU/1/09/529/001; ATC code: A10BX07; CAS number 204656-20-2
  Arms: Liraglutide
Drug: Liraglutide - Placebo — Preparation and labelling of Investigational Medicinal Product:
  Liraglutide - Placebo will be packed and labeled by Novo Nordisk A/S and provided in non-subject specific boxes. Labeling will be in accordance with Annex 13, local law and trial requirements. The examples of labels are not readily available, but will be supplied when received from Novo Nordisk.
  Drug accountability:
  Drug accountability will be cared for by the Department of Clinical Pharmacy of the LUMC. The trial product will be dispensed to each subject as required according to treatment group by the clinical pharmacist. No trial product will be dispensed to any person not enrolled in the trial.
  Other Names: Placebo
  Arms: Liraglutide-placebo

SUMMARY:
The most important cause of mortality amongst DM2 patients is cardiovascular disease. An early finding of cardiovascular disease in DM2 and obesity is diastolic dysfunction. Diastolic dysfunction is an independent predictor of mortality and has been shown to improve in patients on a low calorie diet. The improvement of diastolic function was associated with a reduction in triglyceride accumulation in the heart and liver. A relatively new widely prescribed therapeutic agent for DM2 patients is Liraglutide (Victoza®). Liraglutide is a Glucagon Like Peptide - 1 homologue that improves glucose homeostasis and reduces blood pressure and body weight. Next to the induction of weight loss, which is potentially beneficial for cardiac function, GLP-1 therapy might have a direct advantageous effect on the cardiovascular system. However, the effect of Liraglutide on cardiovascular function has not been investigated yet. The investigators hypothesize that treatment of DM2 patients with Liraglutide is associated with improvement of cardiovascular function and a reduction of triglyceride accumulation in end-organs.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE

   Type 2 diabetes mellitus is an endemic disease associated with obesity and a sedentary lifestyle. In the year 2025 the prevalence of DM2 patients worldwide is expected to be 334 million. In the year 2000 there were an estimated 2,9 million diabetes-related deaths worldwide. Especially cardiovascular disease contributes for a great deal to the high mortality rates. Diabetes patients have a two-fold excess risk for a wide range of vascular diseases, independently of other risk factors, making cardiovascular disease the leading cause of death of diabetes patients. Therefore, treatment of DM2 is focused on the prevention of cardiovascular disease and other diabetes related complications such as retinopathy, neuropathy and nephropathy. Unfortunately, despite lifestyle advises, glucose lowering therapy and co-treatment of other risk factors such as hypertension and dyslipidemia, complication rates remain high. Classical glucose lowering treatment strategies such as sulfonylurea derivatives and insulin ultimately can not control the disease, partly because they participate in the vicious cycle of increasing body weight and insulin resistance. A hopeful new therapeutic agent is the Glucagon Like Peptide -1 analogue Liraglutide. Next to its glucose lowering effect, it reduces body weight resulting in increased insulin sensitivity. The group of GLP-1 analogues are therefore widely prescribed nowadays. However, the effect on the cardiovascular system has not been investigated yet. Since cardiovascular disease is the major threat for the DM2 patient, the effect of this new drug on the cardiovascular system is a very important issue. Interestingly, a cardio-protective effect from Liraglutide can be expected on the basis of both the associated weight loss and because of a direct protective effect on the heart. The investigators hypothesize that treatment with Liraglutide improves cardiac function in DM2 patients. The pathogenesis of cardiovascular disease in DM2 is rather complex and multifactorial. Ultimately most patients develop myocardial infarction and / or heart failure. Often DM2 patients already have subclinical signs of cardiac dysfunction before DM2 is recognized, the main early sign being diastolic dysfunction. Diastolic dysfunction is a strong predictor of mortality. The subclinical characteristics of cardiac dysfunction are highly associated with a condition called the metabolic syndrome. The metabolic syndrome consists of the existence of three out of five of the following risk factors: 1. elevated waist circumference; 2. elevated triglycerides; 3. reduced HDL-C; 4. elevated blood pressure; 5. elevated fasting blood glucose including diabetic-range elevated blood glucose level. With these criteria most patients with diabetes meet the criteria for the metabolic syndrome. A key element in the pathogenesis of the metabolic syndrome might be ectopic fat deposition; the earliest sign of the syndrome being visceral adiposity. Next to visceral adiposity, there is significant deposition of ectopic fat stores in the liver, heart, skeletal muscle and kidney. Triglyceride accumulation in the cardiomyocyte is called myocardial steatosis. Studies performed by our group have proven that caloric restriction results in a reduction in myocardial steatosis and improvement of diastolic function. Hence, myocardial steatosis and associated cardiac dysfunction seem to be reversible as is the case for hepatic steatosis. The putative mechanism of steatosis resulting in cardiac dysfunction is thought to be explained by a phenomenon called lipotoxicity. Altered substrate metabolism and insulin resistance of cardiomyocytes may also play an important role in the pathogenesis of cardiac dysfunction in obesity and DM2. Systemic and cardiac insulin resistance was proven to be associated with increased production of toxic lipids such as diacylglycerol and ceramide. The ultimate treatment for obesity and diabetes related cardiac disease seems to be weight loss. However, lifestyle intervention programs have repeatedly been unsuccessful to have a sustained long term effect. Liraglutide is characterized as a long-acting, human GLP-1 analogue as it shows 97% homology with the amino acid sequence of human GLP-1. The phase 3a program for Liraglutide encompasses five clinical trials in which Liraglutide treatment was studied in each stage of the treatment cascade for type 2 diabetes mellitus. In five studies, Liraglutide was compared directly to standard treatment. The phase 3a clinical development program, included 3,978 exposed patients with DM2, investigated the efficacy and tolerability of Liraglutide 1.2 or 1.8 mg daily (n = 2735) as monotherapy and in combination with various oral antidiabetic drugs. The phase 3a studies showed HBA1C reductions of 1-1.5% and fasting plasma glucose reductions of 0,83 - 2,39 mmol/L. In addition, weight reduction was consistent: Liraglutide 1.8 mg as monotherapy was accompanied by a mean weight loss of 2.5 kg over a 52-week period. A substudy of two phase 3a trials showed that the weight loss caused by Liraglutide, is predominantly caused by a reduction in fat mass; the visceral fat compartment was reduced by 16% from baseline during 26 weeks of Liraglutide 1,2 mg daily. Recent experimental data suggest GLP-1 and its analogues to have direct effects on the heart. In studies on rat heart, the size of an infarct was diminished by more than 50% by an infusion of GLP-1. Post conditioning efficacy of GLP-1 was also demonstrated in an ex vivo rat heart. Exendin-4 was shown to diminish infarct size by approximately 56% and 39%, respectively, in rat global and pig focal models of heart ischemia. The GLP-1 receptor (GLP-1R) is present in the cardiomyocytes as well as in the endothelium and smooth muscle cells of myocardial vasculature. The cell death effector mechanisms targeted by the GLP-1R appear to be mitochondrial permeability transition and apoptosis. Animal studies have suggested myocardial contractility improvement after GLP-1 administration. For instance, dogs with dilated cardiomyopathy treated with GLP-1 for 48 h showed strong improvements in myocardial contractility and cardiac output. GLP-1 infusion was associated with increased myocardial glucose uptake, suggesting ameliorated insulin sensitivity of the cardiomyocytes. In a few small clinical studies, GLP-1 was infused to patients after PCI for approximately 72 h and to patients selected for elective coronary artery bypass grafting from 12 h before to 48 h after the surgery. The latter group showed an improved metabolic profile but no hemodynamic change. In contrast, a left ventricular ejection fraction (LVEF) increase from 29% to 39% was found in the former study, as well as in a study of 12 diabetic, overweight heart failure patients (New York Heart Association class III/IV, LVEF ≤ 40%), given GLP-1 infusion for 5 weeks: at the end of the treatment, these patients showed an increased LVEF, cardiac output, and improved scores in a life quality questionnaire. A number of laboratory studies have suggested a vasorelaxant effect of GLP-1. No pressor effect has been found associated with GLP-1 treatment in studies on diabetic patients. In fact, a decrease of both systolic and diastolic blood pressure values was noted in DM2 patients after an 82-week exenatide trial [33], in a manner correlated to weight loss. Recent experiments (unpublished data) have shown that the GLP-1 analogue exendin - 4 can protect against atherosclerosis and non-alcoholic steatohepatitis (NASH) in APOE 3 - Leiden.CETP mice on a western diet probably due to decreased hepatic CETP expression as well as reduced monocyte recruitment from the circulation to the vessel wall. In addition, hepatic steatosis was improved by a GLP-1 receptor agonist in mice. So far, no dedicated clinical studies have been performed to systematically study the effects of GLP-1 analogues on cardiovascular function. Given the consistency of the results from animal experiments and clinical observations, this area appears ripe for clinical studies. Beneficial effects on cardiovascular endpoints will be crucial to consolidate the therapeutic profile of Liraglutide. Although large scale studies on cardiovascular endpoints are underway, an attractive option is to perform small scale, short-term studies with advanced cardiovascular imaging techniques. Thereby gaining insight in what way GLP-1 therapy affects the cardiovascular system. Advanced cardiovascular magnetic resonance imaging and spectroscopy (MRI/S) enables to assess effects of interventions, in relatively small groups of patients in a limited period of time. As these cardiovascular parameters are strong and clinically relevant predictors of cardiovascular events, measurements of these parameters with MRI/S are worthwhile. Our research group has developed advanced cardiovascular MRI and MRS techniques and algorithms and gained extended experience in the field of DM2 related cardiac function and lipid metabolism.
2. RECRUITMENT AND SCREENING PROCEDURE OF STUDY POPULATION

   Patients will be recruited from the outpatient clinics of the Leiden University Medical Center, general practitioners, local hospitals and by advertisement. Patients own physicists will be asked to point eligible patients to the opportunity of study participation. If interested, patients will be informed by the principal investigator. Patients will be given oral and written explanation about the study. After a consideration time of two weeks, patients are asked to give written acknowledgement of informed consent to participate. Then a medical screening will take place. Screening will be performed after an overnight fast of at least 12 hours. The screening will consist of a medical history, physical examination consisting of measurement of height, body weight, heart rate, blood pressure and examination of thorax and abdomen. Furthermore laboratory tests and rest-ECG will be performed. If the patient is eligible- and willing to participate in the study, and has signed the informed consent, the patient will be included. Informed consent must be obtained before any trial related activities take place. After inclusion in the study protocol, the patient's treating physician and general practitioner will be notified. Although the patients are free to leave the study at any time, it will be attempted to recruit patients who are likely to continue the study to completion.
3. SAMPLE SIZE CALCULATION

   Because of the absence of data on the effects of GLP-1 in DM2 patients without heart failure, it is hard to calculate the sample size needed to detect differences between myocardial function at 26 weeks between active treatment and controls. Clinically relevant differences and standard deviations of two studies were chosen to generate data for the sample size calculation. The data we used to incorporate the precision of MRI assessment of cardiac function was generated by a study performed by our group with pioglitazone vs metformin on cardiac function parameters. To estimate the effect of GLP-1 therapy on cardiac function, we only have data of a pilot study with eight DM2 patients with heart failure. Calculations for diastolic function parameters were based on the "early deceleration peak" and for systolic function on the basis of "ejection fraction". With a power of 90% and alfa = 0.05, groups varying from 9 to 17 patients will be needed. In a comparable trial the drop-out rate was 10%. Taken into consideration that the population studied will have a significant better systolic function than the heart failure patients studied by Sokos et al, differences may be smaller. In conclusion, investigators estimate to be able to detect a clinically relevant, significant result with 90% power and alfa = 0.05 with 25 patients in each group.
4. USE OF CO-INTERVENTION

   Patients should continue to use the oral glucose lowering medicament metformin during the study. For glycaemic control after initiation of the study drug, the current clinical guideline will be followed. Excluded concomitant therapy: thiazolidinediones, other GLP-1 analogues or DPP-IV inhibitors, fibrates, prednisone, cytostatic and antiretroviral therapy.

   Permitted concomitant medication: any other medication required, including SU derivatives, insulin, antihypertensive agents and incidental analgesic and antibiotic therapy. Glycaemic management during study the will be performed as described in appendix 1. To avoid the potential risk of hypoglycaemia, a rigorous monitoring and therapy adjustment schedule will be applied, which will prevent risk of hypoglycemia to a great extent. In addition, patients will be instructed how to recognize and manage a hypo or hyperglycaemic episode. Appropriate individualized adjustments will be made in the unlikely case of a hypo or hyperglycaemic episode. Routine self-measurement of blood glucose by the study participants will be performed once a week. In addition, patients with insulin will be instructed to perform routine self-measurement of blood glucose more frequently when study medication and / or insulin dosage is titrated (see appendix 1).

   Furthermore patients are asked not to change their diet or level of physical activity during the study period and adequate contraception is obligatory for study participation.
5. RANDOMIZATION, BLINDING AND TREATMENT ALLOCATION

   After the medical screening and mutual agreement of participation in the study, patients will be randomized by block randomization, stratified 1:1 for gender and insulin use. A randomization schedule will be prepared by the research pharmacist who is employee at the Department of Clinical Pharmacy. Coded and sealed envelopes for each participant will be kept at the department of Radiology. In case of safety issues, the sealed envelopes are readily available to the principal investigator and project leader. In case of a serious adverse event - or a medical emergency requiring knowledge of the study medication - the randomization code will be broken. In order to ensure that in medical emergencies, the study participation of the patient is apparent, each patient will receive a patient file in the electronic patient registry. In this personal file, the study number of the patient including the procedure for deblinding and notification of the investigators will be mentioned. When the whole study is completed the randomization list will be provided to the principle investigator by the pharmacist.
6. STUDY PROCEDURES

   Withdrawal of individual subjects: Patients can leave the study at any time for any reason if they wish to do so without any consequences. The responsible investigator can also withdraw a subject if continuing participation is in his opinion deleterious for the subject's well being. Patients can also be withdrawn in case of protocol violations and non-compliance. When a subject withdraws from the study, a medical examination will be performed. In case of withdrawal because of a severe or serious adverse event, appropriate laboratory tests or other special examinations will be performed. Finally patients can be withdrawn from study participation if an incidental finding at the MRI examination - for example a malignancy - influences the ratio of justification versus risks / benefits.

   Specific criteria for withdrawal: not applicable

   Replacement of individual subjects after withdrawal: Patients will not be replaced after withdrawal.

   Follow-up of subjects withdrawn from treatment: Follow-up of patients after withdrawal will be done by the treating physicist (general practitioner in most cases). Immediately after study withdrawal, the treating physicist will be updated on the patient's condition and laboratory results and whether the patient was in the control group or intervention group.

   Premature termination of the study: In case of the incidence of three serious adverse events, the study will be terminated prematurely and an independent committee will be asked to investigate the safety of the trial. Furthermore, the investigators will prematurely terminate the study when the number of subjects withdrawn from the study exceeds the number used for sample size calculation, i.e. 16 individuals in total.
7. ADVERSE EVENTS, SERIOUS ADVERSE EVENTS and SUSPECTED UNEXPECTED SERIOUS ADVERSE REACTIONS

Adverse events (AEs):

Adverse events are defined as any undesirable experience occurring to a subject during a clinical trial, whether or not considered related to the used medication or the infused drugs. All adverse events reported spontaneously by the subject or observed by the investigator or his/her staff will be recorded on the adverse event data collection form. The intensity of these adverse events will be graded by the investigator as follows:

* Mild: Discomfort noted but no disruption of normal daily activity
* Moderate: Discomfort sufficient to reduce or affect normal daily activity
* Severe: Inability to work or perform daily activity All adverse events will be actively queried by asking the question: "Have you had any complaints since the last time we talked/met?" at all visits. All adverse events will be followed until they have abated, or until a stable situation has been reached. Depending on the event, follow up may require additional tests or medical procedures as indicated.

The chronicity of the event will be classified by the investigator on a three-item scale as defined below:

* Single occasion: Single event with limited duration
* Intermittent: Several episodes of an event, each of limited duration
* Persistent: Event that remains indefinitely For each adverse event, the relationship to the used medication or infused drug (definite, probable, possible, unknown, definitively not) as judged by the investigator, will be recorded, as well as any actions undertaken in relation to the adverse event, will be recorded. The occurrence of an adverse event that is fatal, life-threatening, disabling or requires in-patient hospitalization, or causes congenital anomaly, will be described according to CHMP guidelines as (suspected) "serious" adverse events and will be notified in writing to the Medical Ethics Committee.

Furthermore, the investigators will copy Novo Nordisk when expediting SARs and SUSARs to competent authorities and will report all SARs related to Novo Nordisk product to Novo Nordisk. The submission to Novo Nordisk must however be within day 15 from the investigator getting knowledge about a valid case no matter local timelines for reporting to the authorities. All pregnancies in trial patients occurring during use of a Novo Nordisk product must be reported to Novo Nordisk.

Serious Adverse Events (SAEs):

A serious adverse event is any untoward medical occurrence or effect that at any dose:

* results in death;
* is life threatening (at the time of the event);
* requires hospitalization or prolongation of existing inpatients' hospitalization;
* results in persistent or significant disability or incapacity;
* is a congenital anomaly or birth defect;
* Any other important medical event that may not result in death, be life threatening, or require hospitalization, may be considered a serious adverse experience when, based upon appropriate medical judgement, the event may jeopardize the subject or may require an intervention to prevent one of the outcomes listed above.

The sponsor will report the SAEs to the accredited METC that approved the protocol, within 15 days after the sponsor has first knowledge of the serious adverse reactions.

SAEs that result in death or are life threatening should be reported expedited. The expedited reporting will occur not later than 7 days after the responsible investigator has first knowledge of the adverse reaction. This is for a preliminary report with another 8 days for completion of the report.

Suspected Unexpected Serious Adverse Reactions (SUSARs):

Unexpected adverse reactions are SUSARs if the following three conditions are met:

1. the event must be serious
2. there must be a certain degree of probability that the event is a harmful and an undesirable reaction to the medicinal product under investigation, regardless of the administered dose;
3. the adverse reaction must be unexpected, that is to say, the nature and severity of the adverse reaction are not in agreement with the product information as recorded in:

   * Summary of Product Characteristics (SPC) for an authorized medicinal product;
   * Investigator's Brochure for an unauthorized medicinal product. The sponsor will report expedited all SUSARs to the competent authorities in other Member States, according to the requirements of the Member States.

The expedited reporting will occur not later than 15 days after the sponsor has first knowledge of the adverse reactions. For fatal or life threatening cases the term will be maximal 7 days for a preliminary report with another 8 days for completion of the report.

SAEs need to be reported till end of study within the Netherlands, as defined in the protocol

8. STATISTICAL ANALYSIS

Primary and secondary study parameters:

The study endpoints will be analyzed according to intention-to-treat principles. All endpoint parameters are continuous variables. Data will be calculated as mean SD, median (percentile range) according to nature and distribution of the variable. Within group changes from baseline will be tested with independent paired t-test or Wilcoxon signed-rank test. Between group differences will be compared after 26 weeks between Liraglutide and control. The endpoints will be analyzed using a linear regression model, with gender, age, BMI and HBA1C as covariates. For the covariates age, BMI and HbA1c in the primary analysis the baseline value will be used. The data set for the primary analysis will include data from all subjects with at least one post-baseline measurement. Analysis will be performed with SPSS. A 2-sided significance level of p < 0.05 will be applied.

9 REGULATION STATEMENT

The study will be conducted according to the principles of the "Declaration of Helsinki" (as amended in Tokyo, Venice and Hong Kong, Somerset West and Edinburgh) and in accordance with the Guideline for Good Clinical Practice (CPMP/ICH/135/95 - 17th July 1996).

10. ADMINISTRATIVE ASPECTS, MONITORING AND PUBLICATION

Handling and storage of data and documents:

Study participants are provided a study name of the letter "MV" followed by the number of enrollment (1-50). The study name is coupled to a randomly chosen seven - digit study number. The study number will be used to register the participant in the Electronic Patient Registry of the LUMC. This file will be used as the general patient record, as well as collection of routine laboratory measurements needed for clinical and study treatment. The MRI images will be filed under this registry so that anonymity will be safeguarded. The subject identification code list will be stored by the principal investigator and will only be accessible by the principal investigator and project leader. The data extracted from the study file in the Electronic Patient Registry and from the MRI images will be saved in an SPSS file. From this file the true identity of the study participants can not be discovered. The data will be stored for fifteen years. The blood samples will be frozen and stored anonymously using the above mentioned study name and study number. For ad hoc laboratory tests of inflammatory, endocrine and other biomarkers, blood samples will be kept for a maximum period of three years. The blood samples are solely accessible by the investigator team.

In order to ensure that in medical emergencies, the study participation of the patient is apparent, each patient will receive a patient file in the electronic patient registry. In this personal file, the investigator will mention the study number of the patient including the procedure for de-blinding and notification of the investigators. In this file, the signed Informed Consent form of the patient will be stored.

Public disclosure and publication policy: The data analysis will be performed by the investigators. Novo Nordisk has no role in data analysis and / or publication of the results of the trial in peer reviewed papers. The results of the study will be submitted to peer reviewed papers, also in case the hypothesis has not been proven.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age > 18 years and < 70 years
* BMI > 25 kg/m2
* DM2 treated with metformin, metformin + SU derivative, metformin + SU derivative + insulin, or metformin + insulin for at least 3 months in the maximum tolerable dosage
* HbA1c ≥7% and ≤ 10.0 %
* EGFR > 60 ml/min
* Normal sitting blood pressure < 150/85 mm Hg and stable for at least one month

Exclusion Criteria:

* Use of thiazolidinediones (TZD), GLP-1 analogues, DPP-IV inhibitors, fibrates, prednisone, cytostatic or antiretroviral therapy within 6 months prior to the study
* Hereditary lipoprotein disease
* Psychiatric disorders and / or use of antipsychotic or antidepressant drugs at present or in the past
* Hepatic disease (AST/ALT > 2 times reference values)
* Endocrine disease other than diabetes mellitus type 2
* History or presence of cardiovascular disease
* Any significant chronic disease (e.g. inflammatory bowel disease)
* Any significant abnormal laboratory results found during the medical screening procedure
* Gastrointestinal surgery (e.g. gastric bypass)
* Pregnant woman or a woman who is breast-feeding
* Female of child-bearing potential intending to become pregnant or is not using adequate contraceptive methods while sexually active
* Allergy to intravenous contrast
* Known or suspected hypersensitivity to trial products or related products
* Chronic pancreatitis or previous acute pancreatitis
* Personal history or family history of medullary thyroid carcinoma or personal history of multiple endocrine neoplasia type 2
* Claustrophobia
* Metal implants or other contraindications for MRI
* Recent participation in other research projects within the last 3 months or participation in 2 or more projects in one year

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Stroke volume | 0 and 26 weeks
  Change from baseline in ml: difference between groups
Ejection Fraction | 0 and 26 weeks
  Change from baseline in percentage: difference between groups
Cardiac output | 0 and 26 weeks
  Change from baseline in L/min: difference between groups
Cardiac index | 0 and 26 weeks
  Change from baseline in L/min/m2: difference between groups
Peak ejection rate | 0 and 26 weeks
  Change from baseline in ml end-diastolic volume/sec: difference between groups
Early peak filling rate | 0 and 26 weeks
  Change from baseline in ml end-diastolic volume/sec: difference between groups
Early deceleration peak | 0 and 26 weeks
  Change from baseline in ml/sec: difference between groups
Atrial peak filling rate | 0 and 26 weeks
  Change from baseline in ml/sec: difference between groups
Early deceleration peak / Atrial peak filling rate (E/A ratio) | 0 and 26 weeks
  Change from baseline of the ratio: difference between groups
Peak mitral annulus longitudinal motion | 0 and 26 weeks
  Change from baseline in cm/sec: difference between groups
Left ventricular filling pressure (= early peak filling rate / peak mitral annulus longitudinal motion) | 0 and 26 weeks
  Change from baseline in mmHg: difference between groups

SECONDARY OUTCOMES:
Aorta and carotid vessel wall imaging | 0 and 26 weeks
  Change from baseline of total vessel wall area in mm2: difference between groups
Aorta and carotid vessel wall imaging | 0 and 26 weeks
  Change from baseline of average vessel wall thickness in mm: difference between groups
Aorta and carotid vessel wall imaging | 0 and 26 weeks
  Change from baseline of a minimum vessel wall thickness in mm: difference between groups
Aorta and carotid vessel wall imaging | 0 and 26 weeks
  Change from baseline of maximum vessel wall thickness in mm: difference between groups
Aorta and carotid vessel wall imaging | 0 and 26 weeks
  Change from baseline of vascular distensibility (pulse wave velocity): difference between groups
Adipose tissue distribution | 0 and 26 weeks
  Change from baseline of the ratio subcutaneous fat / visceral abdominal fat: difference between groups
Total body fat | 0 and 26 weeks
  Change from baseline of total fat volume in ml: difference between groups
Epicardial fat volume | 0 and 26 weeks
  Change from baseline in cm3: difference between groups
Magnetic Resonance Spectroscopy of the heart | 0 and 26 weeks
  Change from baseline in percentage: difference between groups
Magnetic Resonance Spectroscopy of the liver | 0 and 26 weeks
  Change from baseline in percentage: difference between groups
Magnetic Resonance Spectroscopy of the kidney | 0 and 26 weeks
  Change from baseline in percentage: difference between groups
HBA1C | 0,8, 12, 16 and 26 weeks
  Measurements will be used to guide therapeutic management
  The outcome measure glycemic control will be based on the average HBA1C level of all measurements and regards: difference between groups.
Fasting blood glucose level | 0, 4, 8, 12, 16, 20, 26 weeks
  Fasting blood glucose levels will be used to guide therapeutic management and for safety reasons.
  Outcome measure: the difference between groups of the average of all measurements.
Myocardial T1 - mapping | 0 and 26 weeks
  Change from baseline of myocardial T1 - values before and after contrast: difference between groups

OTHER OUTCOMES:
Anthropometric measurements | 0, 4, 8, 12, 16, 20, 26 weeks
  Length, body weight and calculated BMI.
  Outcome measure: Change from baseline in kg (body weight) or kg/m2 (BMI): difference between groups
Waist / hip ratio | 0, 4, 8, 12, 16, 20, 26 weeks
  Waist circumference divided by hip circumference.
  Outcome measure: change from baseline: difference between groups
Systolic blood pressure | 0, 4, 8, 12, 16, 20, 26 weeks
  Measurements for routine clinical management
  Outcome measure: change from baseline in mmHg: difference between groups
Diastolic blood pressure | 0, 4, 8, 12, 16, 20, 26 weeks
  Measurements for routine clinical management
  Outcome measure: change from baseline in mmHg: difference between groups
Resting Energy Expenditure | 0, 4, 12, 26 weeks
  Change from baseline: difference between groups
  Measurement with indirect calorimetry (Jaeger, OxyconPro)
Immunological analysis | 0, 26 weeks
  Fluorescence-Activated Cell Sorting (FACS).
  Change from baseline: difference between groups.
Immunological analysis | 0, 26 weeks
  Peripheral Blood Mononuclear Cell isolation to analyze immunological activation and status of subjects. Both quantification of white blood cells (T-cells, B-cells, macrophages) and functional analysis will be performed.
  Change from baseline: difference between groups
Fasting insulin level | 0 and 26 weeks
  Change from baseline: difference between groups
Leptin | 0 and 26 weeks
  Change from baseline: difference between groups
Glucagon | 0 and 26 weeks
  Change from baseline: difference between groups
Adiponectin | 0 and 26 weeks
  Change from baseline: difference between groups
CETP | 0, 4, 12 and 26 weeks
  Cholesteryl ester transfer protein
  Change from baseline: difference between groups
High Sensitive C Reactive Protein | 0, 4, 12 and 26 weeks
  Change from baseline: difference between groups
Free Fatty Acids | 0, 4, 12 and 26 weeks
  Change from baseline: difference between groups
Cholesterol level (total, HDL and LDL) | 0, 4, 12 and 26 weeks
  Change from baseline: difference between groups
Liver function tests (ALT, AST, AF, GGT) | 0, 4, 12 and 26 weeks
  Change from baseline: difference between groups
Triglycerides | 0, 4 , 12 and 26 weeks
  Change from baseline: difference between groups
QUICKI | 0 and 26 weeks
  Quantitative Insulin Sensitivity Check Index
  Change from baseline: difference between groups
Albuminuria | 0 and 26 weeks
  Change from baseline of urinary albumin / creatinine ration: difference between groups
Immunological analysis | 0 and 26 weeks
  Immunological status as assessed by RNA profiling. Change from baseline: difference between groups
Metabolomics | 0 and 26 weeks
  Metabolomics in urine and blood sample. Change from baseline: difference between groups
Insulin dose | 0 and 26 weeks
  Total daily dose (units) of insulin. Change from baseline: difference between groups
Hypoglycaemic episodes | Between week 0 and 26
  Number of grade 1, 2 and 3 hypoglycaemic episodes as detected with self measurement by participants. Comparison between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Maurice B Bizino, MD, Principal Investigator — Leiden University Medical Center; Jan WA Smit, MD PhD, Study Chair — University Nijmegen Medical Centre; Hildo J Lamb, MD PhD, Study Director — Leiden University Medical Center; Albert de Roos, MD PhD, Study Chair — Leiden University Medical Center; Ingrid M Jazet, MD PhD, Study Chair — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Roglic G, Unwin N, Bennett PH, Mathers C, Tuomilehto J, Nag S, Connolly V, King H. The burden of mortality attributable to diabetes: realistic estimates for the year 2000. Diabetes Care. 2005 Sep;28(9):2130-5. doi: 10.2337/diacare.28.9.2130. PMID 16123478
- [Background] Emerging Risk Factors Collaboration; Sarwar N, Gao P, Seshasai SR, Gobin R, Kaptoge S, Di Angelantonio E, Ingelsson E, Lawlor DA, Selvin E, Stampfer M, Stehouwer CD, Lewington S, Pennells L, Thompson A, Sattar N, White IR, Ray KK, Danesh J. Diabetes mellitus, fasting blood glucose concentration, and risk of vascular disease: a collaborative meta-analysis of 102 prospective studies. Lancet. 2010 Jun 26;375(9733):2215-22. doi: 10.1016/S0140-6736(10)60484-9. PMID 20609967
- [Background] Abi Khalil C, Roussel R, Mohammedi K, Danchin N, Marre M. Cause-specific mortality in diabetes: recent changes in trend mortality. Eur J Prev Cardiol. 2012 Jun;19(3):374-81. doi: 10.1177/1741826711409324. PMID 22991697
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] van der Meer RW, Lamb HJ, Smit JW, de Roos A. MR imaging evaluation of cardiovascular risk in metabolic syndrome. Radiology. 2012 Jul;264(1):21-37. doi: 10.1148/radiol.12110772. PMID 22723560
- [Background] Celentano A, Vaccaro O, Tammaro P, Galderisi M, Crivaro M, Oliviero M, Imperatore G, Palmieri V, Iovino V, Riccardi G, et al. Early abnormalities of cardiac function in non-insulin-dependent diabetes mellitus and impaired glucose tolerance. Am J Cardiol. 1995 Dec 1;76(16):1173-6. doi: 10.1016/s0002-9149(99)80330-0. PMID 7484905
- [Background] Bella JN, Palmieri V, Roman MJ, Liu JE, Welty TK, Lee ET, Fabsitz RR, Howard BV, Devereux RB. Mitral ratio of peak early to late diastolic filling velocity as a predictor of mortality in middle-aged and elderly adults: the Strong Heart Study. Circulation. 2002 Apr 23;105(16):1928-33. doi: 10.1161/01.cir.0000015076.37047.d9. PMID 11997279
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] Machann J, Haring H, Schick F, Stumvoll M. Intramyocellular lipids and insulin resistance. Diabetes Obes Metab. 2004 Jul;6(4):239-48. doi: 10.1111/j.1462-8902.2004.00339.x. PMID 15171747
- [Background] McGavock JM, Lingvay I, Zib I, Tillery T, Salas N, Unger R, Levine BD, Raskin P, Victor RG, Szczepaniak LS. Cardiac steatosis in diabetes mellitus: a 1H-magnetic resonance spectroscopy study. Circulation. 2007 Sep 4;116(10):1170-5. doi: 10.1161/CIRCULATIONAHA.106.645614. Epub 2007 Aug 13. PMID 17698735
- [Background] Thomas EL, Hamilton G, Patel N, O'Dwyer R, Dore CJ, Goldin RD, Bell JD, Taylor-Robinson SD. Hepatic triglyceride content and its relation to body adiposity: a magnetic resonance imaging and proton magnetic resonance spectroscopy study. Gut. 2005 Jan;54(1):122-7. doi: 10.1136/gut.2003.036566. PMID 15591516
- [Background] Despres JP. Body fat distribution and risk of cardiovascular disease: an update. Circulation. 2012 Sep 4;126(10):1301-13. doi: 10.1161/CIRCULATIONAHA.111.067264. No abstract available. PMID 22949540
- [Background] Hammer S, Snel M, Lamb HJ, Jazet IM, van der Meer RW, Pijl H, Meinders EA, Romijn JA, de Roos A, Smit JW. Prolonged caloric restriction in obese patients with type 2 diabetes mellitus decreases myocardial triglyceride content and improves myocardial function. J Am Coll Cardiol. 2008 Sep 16;52(12):1006-12. doi: 10.1016/j.jacc.2008.04.068. PMID 18786482
- [Background] Hammer S, van der Meer RW, Lamb HJ, Schar M, de Roos A, Smit JW, Romijn JA. Progressive caloric restriction induces dose-dependent changes in myocardial triglyceride content and diastolic function in healthy men. J Clin Endocrinol Metab. 2008 Feb;93(2):497-503. doi: 10.1210/jc.2007-2015. Epub 2007 Nov 20. PMID 18029455
- [Background] Chokshi A, Drosatos K, Cheema FH, Ji R, Khawaja T, Yu S, Kato T, Khan R, Takayama H, Knoll R, Milting H, Chung CS, Jorde U, Naka Y, Mancini DM, Goldberg IJ, Schulze PC. Ventricular assist device implantation corrects myocardial lipotoxicity, reverses insulin resistance, and normalizes cardiac metabolism in patients with advanced heart failure. Circulation. 2012 Jun 12;125(23):2844-53. doi: 10.1161/CIRCULATIONAHA.111.060889. Epub 2012 May 14. PMID 22586279
- [Background] Schaffer JE. Lipotoxicity: when tissues overeat. Curr Opin Lipidol. 2003 Jun;14(3):281-7. doi: 10.1097/00041433-200306000-00008. PMID 12840659
- [Background] Hensrud DD. Dietary treatment and long-term weight loss and maintenance in type 2 diabetes. Obes Res. 2001 Nov;9 Suppl 4:348S-353S. doi: 10.1038/oby.2001.141. PMID 11707564
- [Background] Jendle J, Nauck MA, Matthews DR, Frid A, Hermansen K, During M, Zdravkovic M, Strauss BJ, Garber AJ; LEAD-2 and LEAD-3 Study Groups. Weight loss with liraglutide, a once-daily human glucagon-like peptide-1 analogue for type 2 diabetes treatment as monotherapy or added to metformin, is primarily as a result of a reduction in fat tissue. Diabetes Obes Metab. 2009 Dec;11(12):1163-72. doi: 10.1111/j.1463-1326.2009.01158.x. PMID 19930006
- [Background] Bose AK, Mocanu MM, Carr RD, Yellon DM. Glucagon like peptide-1 is protective against myocardial ischemia/reperfusion injury when given either as a preconditioning mimetic or at reperfusion in an isolated rat heart model. Cardiovasc Drugs Ther. 2005 Jan;19(1):9-11. doi: 10.1007/s10557-005-6892-4. No abstract available. PMID 15883751
- [Background] Ossum A, van Deurs U, Engstrom T, Jensen JS, Treiman M. The cardioprotective and inotropic components of the postconditioning effects of GLP-1 and GLP-1(9-36)a in an isolated rat heart. Pharmacol Res. 2009 Nov;60(5):411-7. doi: 10.1016/j.phrs.2009.06.004. Epub 2009 Jun 18. PMID 19540343
- [Background] Sonne DP, Engstrom T, Treiman M. Protective effects of GLP-1 analogues exendin-4 and GLP-1(9-36) amide against ischemia-reperfusion injury in rat heart. Regul Pept. 2008 Feb 7;146(1-3):243-9. doi: 10.1016/j.regpep.2007.10.001. Epub 2007 Oct 13. PMID 17976835
- [Background] Timmers L, Henriques JP, de Kleijn DP, Devries JH, Kemperman H, Steendijk P, Verlaan CW, Kerver M, Piek JJ, Doevendans PA, Pasterkamp G, Hoefer IE. Exenatide reduces infarct size and improves cardiac function in a porcine model of ischemia and reperfusion injury. J Am Coll Cardiol. 2009 Feb 10;53(6):501-10. doi: 10.1016/j.jacc.2008.10.033. PMID 19195607
- [Background] Ban K, Noyan-Ashraf MH, Hoefer J, Bolz SS, Drucker DJ, Husain M. Cardioprotective and vasodilatory actions of glucagon-like peptide 1 receptor are mediated through both glucagon-like peptide 1 receptor-dependent and -independent pathways. Circulation. 2008 May 6;117(18):2340-50. doi: 10.1161/CIRCULATIONAHA.107.739938. Epub 2008 Apr 21. PMID 18427132
- [Background] Nikolaidis LA, Elahi D, Hentosz T, Doverspike A, Huerbin R, Zourelias L, Stolarski C, Shen YT, Shannon RP. Recombinant glucagon-like peptide-1 increases myocardial glucose uptake and improves left ventricular performance in conscious dogs with pacing-induced dilated cardiomyopathy. Circulation. 2004 Aug 24;110(8):955-61. doi: 10.1161/01.CIR.0000139339.85840.DD. Epub 2004 Aug 16. PMID 15313949
- [Background] Nikolaidis LA, Mankad S, Sokos GG, Miske G, Shah A, Elahi D, Shannon RP. Effects of glucagon-like peptide-1 in patients with acute myocardial infarction and left ventricular dysfunction after successful reperfusion. Circulation. 2004 Mar 2;109(8):962-5. doi: 10.1161/01.CIR.0000120505.91348.58. Epub 2004 Feb 23. PMID 14981009
- [Background] Sokos GG, Bolukoglu H, German J, Hentosz T, Magovern GJ Jr, Maher TD, Dean DA, Bailey SH, Marrone G, Benckart DH, Elahi D, Shannon RP. Effect of glucagon-like peptide-1 (GLP-1) on glycemic control and left ventricular function in patients undergoing coronary artery bypass grafting. Am J Cardiol. 2007 Sep 1;100(5):824-9. doi: 10.1016/j.amjcard.2007.05.022. Epub 2007 Jun 14. PMID 17719327
- [Background] Sokos GG, Nikolaidis LA, Mankad S, Elahi D, Shannon RP. Glucagon-like peptide-1 infusion improves left ventricular ejection fraction and functional status in patients with chronic heart failure. J Card Fail. 2006 Dec;12(9):694-9. doi: 10.1016/j.cardfail.2006.08.211. PMID 17174230
- [Background] Green BD, Hand KV, Dougan JE, McDonnell BM, Cassidy RS, Grieve DJ. GLP-1 and related peptides cause concentration-dependent relaxation of rat aorta through a pathway involving KATP and cAMP. Arch Biochem Biophys. 2008 Oct 15;478(2):136-42. doi: 10.1016/j.abb.2008.08.001. Epub 2008 Aug 7. PMID 18708025
- [Background] Nystrom T, Gonon AT, Sjoholm A, Pernow J. Glucagon-like peptide-1 relaxes rat conduit arteries via an endothelium-independent mechanism. Regul Pept. 2005 Feb 15;125(1-3):173-7. doi: 10.1016/j.regpep.2004.08.024. PMID 15582729
- [Background] Nystrom T, Gutniak MK, Zhang Q, Zhang F, Holst JJ, Ahren B, Sjoholm A. Effects of glucagon-like peptide-1 on endothelial function in type 2 diabetes patients with stable coronary artery disease. Am J Physiol Endocrinol Metab. 2004 Dec;287(6):E1209-15. doi: 10.1152/ajpendo.00237.2004. Epub 2004 Sep 7. PMID 15353407
- [Background] Zander M, Madsbad S, Madsen JL, Holst JJ. Effect of 6-week course of glucagon-like peptide 1 on glycaemic control, insulin sensitivity, and beta-cell function in type 2 diabetes: a parallel-group study. Lancet. 2002 Mar 9;359(9309):824-30. doi: 10.1016/S0140-6736(02)07952-7. PMID 11897280
- [Background] Blonde L, Klein EJ, Han J, Zhang B, Mac SM, Poon TH, Taylor KL, Trautmann ME, Kim DD, Kendall DM. Interim analysis of the effects of exenatide treatment on A1C, weight and cardiovascular risk factors over 82 weeks in 314 overweight patients with type 2 diabetes. Diabetes Obes Metab. 2006 Jul;8(4):436-47. doi: 10.1111/j.1463-1326.2006.00602.x. PMID 16776751
- [Background] Ding X, Saxena NK, Lin S, Gupta NA, Anania FA. Exendin-4, a glucagon-like protein-1 (GLP-1) receptor agonist, reverses hepatic steatosis in ob/ob mice. Hepatology. 2006 Jan;43(1):173-81. doi: 10.1002/hep.21006. PMID 16374859
- [Background] Diamant M, Lamb HJ, Groeneveld Y, Endert EL, Smit JW, Bax JJ, Romijn JA, de Roos A, Radder JK. Diastolic dysfunction is associated with altered myocardial metabolism in asymptomatic normotensive patients with well-controlled type 2 diabetes mellitus. J Am Coll Cardiol. 2003 Jul 16;42(2):328-35. doi: 10.1016/s0735-1097(03)00625-9. PMID 12875772
- [Background] Hammer S, van der Meer RW, Lamb HJ, de Boer HH, Bax JJ, de Roos A, Romijn JA, Smit JW. Short-term flexibility of myocardial triglycerides and diastolic function in patients with type 2 diabetes mellitus. Am J Physiol Endocrinol Metab. 2008 Sep;295(3):E714-8. doi: 10.1152/ajpendo.90413.2008. Epub 2008 Jul 15. PMID 18628354
- [Background] Jonker JT, Lamb HJ, van der Meer RW, Rijzewijk LJ, Menting LJ, Diamant M, Bax JJ, de Roos A, Romijn JA, Smit JW. Pioglitazone compared with metformin increases pericardial fat volume in patients with type 2 diabetes mellitus. J Clin Endocrinol Metab. 2010 Jan;95(1):456-60. doi: 10.1210/jc.2009-1441. Epub 2009 Nov 13. PMID 19915017
- [Background] Rijzewijk LJ, van der Meer RW, Lamb HJ, de Jong HW, Lubberink M, Romijn JA, Bax JJ, de Roos A, Twisk JW, Heine RJ, Lammertsma AA, Smit JW, Diamant M. Altered myocardial substrate metabolism and decreased diastolic function in nonischemic human diabetic cardiomyopathy: studies with cardiac positron emission tomography and magnetic resonance imaging. J Am Coll Cardiol. 2009 Oct 13;54(16):1524-32. doi: 10.1016/j.jacc.2009.04.074. PMID 19815124
- [Background] van der Meer RW, Doornbos J, Kozerke S, Schar M, Bax JJ, Hammer S, Smit JW, Romijn JA, Diamant M, Rijzewijk LJ, de Roos A, Lamb HJ. Metabolic imaging of myocardial triglyceride content: reproducibility of 1H MR spectroscopy with respiratory navigator gating in volunteers. Radiology. 2007 Oct;245(1):251-7. doi: 10.1148/radiol.2451061904. PMID 17885193
- [Background] van der Meer RW, Hammer S, Lamb HJ, Frolich M, Diamant M, Rijzewijk LJ, de Roos A, Romijn JA, Smit JW. Effects of short-term high-fat, high-energy diet on hepatic and myocardial triglyceride content in healthy men. J Clin Endocrinol Metab. 2008 Jul;93(7):2702-8. doi: 10.1210/jc.2007-2524. Epub 2008 Apr 22. PMID 18430773
- [Background] van der Meer RW, Rijzewijk LJ, de Jong HW, Lamb HJ, Lubberink M, Romijn JA, Bax JJ, de Roos A, Kamp O, Paulus WJ, Heine RJ, Lammertsma AA, Smit JW, Diamant M. Pioglitazone improves cardiac function and alters myocardial substrate metabolism without affecting cardiac triglyceride accumulation and high-energy phosphate metabolism in patients with well-controlled type 2 diabetes mellitus. Circulation. 2009 Apr 21;119(15):2069-77. doi: 10.1161/CIRCULATIONAHA.108.803916. Epub 2009 Apr 6. PMID 19349323
- [Background] Garber A, Henry R, Ratner R, Garcia-Hernandez PA, Rodriguez-Pattzi H, Olvera-Alvarez I, Hale PM, Zdravkovic M, Bode B; LEAD-3 (Mono) Study Group. Liraglutide versus glimepiride monotherapy for type 2 diabetes (LEAD-3 Mono): a randomised, 52-week, phase III, double-blind, parallel-treatment trial. Lancet. 2009 Feb 7;373(9662):473-81. doi: 10.1016/S0140-6736(08)61246-5. Epub 2008 Sep 24. PMID 18819705
- [Background] Marre M, Shaw J, Brandle M, Bebakar WM, Kamaruddin NA, Strand J, Zdravkovic M, Le Thi TD, Colagiuri S; LEAD-1 SU study group. Liraglutide, a once-daily human GLP-1 analogue, added to a sulphonylurea over 26 weeks produces greater improvements in glycaemic and weight control compared with adding rosiglitazone or placebo in subjects with Type 2 diabetes (LEAD-1 SU). Diabet Med. 2009 Mar;26(3):268-78. doi: 10.1111/j.1464-5491.2009.02666.x. PMID 19317822
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Hoekx CA, Martinez-Tellez B, Straat ME, Bizino MB, van Eyk HJ, Lamb HJ, Smit JWA, Jazet IM, Nahon KJ, Janssen LGM, Rensen PCN, Boon MR. Circulating FGF21 is lower in South Asians compared with Europids with type 2 diabetes mellitus. Endocr Connect. 2025 Jan 6;14(2):e240362. doi: 10.1530/EC-24-0362. Print 2025 Feb 1. PMID 39641307
- [Derived] Straat ME, Martinez-Tellez B, van Eyk HJ, Bizino MB, van Veen S, Vianello E, Stienstra R, Ottenhoff THM, Lamb HJ, Smit JWA, Jazet IM, Rensen PCN, Boon MR. Differences in Inflammatory Pathways Between Dutch South Asians vs Dutch Europids With Type 2 Diabetes. J Clin Endocrinol Metab. 2023 Mar 10;108(4):931-940. doi: 10.1210/clinem/dgac598. PMID 36262060
- [Derived] Dekkers IA, Bizino MB, Paiman EHM, Smit JW, Jazet IM, de Vries APJ, Lamb HJ. The Effect of Glycemic Control on Renal Triglyceride Content Assessed by Proton Spectroscopy in Patients With Type 2 Diabetes Mellitus: A Single-Center Parallel-Group Trial. J Ren Nutr. 2021 Nov;31(6):611-619. doi: 10.1053/j.jrn.2020.09.006. Epub 2020 Dec 5. PMID 33293204
- [Derived] van Eyk HJ, Paiman EHM, Bizino MB, IJzermans SL, Kleiburg F, Boers TGW, Rappel EJ, Burakiewicz J, Kan HE, Smit JWA, Lamb HJ, Jazet IM, Rensen PCN. Liraglutide decreases energy expenditure and does not affect the fat fraction of supraclavicular brown adipose tissue in patients with type 2 diabetes. Nutr Metab Cardiovasc Dis. 2020 Apr 12;30(4):616-624. doi: 10.1016/j.numecd.2019.12.005. Epub 2019 Dec 13. PMID 32127340
- [Derived] Bizino MB, Jazet IM, de Heer P, van Eyk HJ, Dekkers IA, Rensen PCN, Paiman EHM, Lamb HJ, Smit JW. Placebo-controlled randomised trial with liraglutide on magnetic resonance endpoints in individuals with type 2 diabetes: a pre-specified secondary study on ectopic fat accumulation. Diabetologia. 2020 Jan;63(1):65-74. doi: 10.1007/s00125-019-05021-6. Epub 2019 Nov 5. PMID 31690988
- [Derived] van Eyk HJ, Blauw LL, Bizino MB, Wang Y, van Dijk KW, de Mutsert R, Smit JWA, Lamb HJ, Jazet IM, Rensen PCN. Hepatic triglyceride content does not affect circulating CETP: lessons from a liraglutide intervention trial and a population-based cohort. Sci Rep. 2019 Jul 10;9(1):9996. doi: 10.1038/s41598-019-45593-2. PMID 31292457
- [Derived] Bizino MB, Jazet IM, Westenberg JJM, van Eyk HJ, Paiman EHM, Smit JWA, Lamb HJ. Effect of liraglutide on cardiac function in patients with type 2 diabetes mellitus: randomized placebo-controlled trial. Cardiovasc Diabetol. 2019 Apr 30;18(1):55. doi: 10.1186/s12933-019-0857-6. PMID 31039778